CLINICAL TRIAL: NCT05939609
Title: Effect of Hamstring-targeted Physiotherapy on Low Back Pain and Muscle Viscoelastic Properties in Elite Adolescent Rowers: A Single-blind Randomized Controlled Trial
Brief Title: Hamstring Viscoelasticity and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Yeditepe University (Other)
Responsible Party: Principal Investigator, Onur Atakan Sekibağ, Principal Investigator, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AtakanS
Record Dates: First submitted 2023-07-01; First posted 2023-07-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain; Athletic Injuries
Keywords: Ballistic Stretching; Athletic Tape; Eccentric Exercise; Low Back Pain; Athletic Performance
MeSH Terms: conditions — Low Back Pain; Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be divided into three groups with equal numbers by computer randomization method.
Who Masked: Outcomes Assessor
Masking Description: The investigator administering the treatment and the investigator performing the evaluations will be different. The evaluator will not know about the interventions that the participants received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ballistic Stretching Exercise (Active Comparator): Athletes will be asked to reach the floor by leaning over in the standing posture without knee flexion. When they feel the tension in hamstring muscle groups, athletes will be requested to make small rebounding motion at degrees between 3°-5° for half a minute.
  Interventions: Other: Ballistic Stretching Exercise
- Extender Exercise (Active Comparator): Athletes will lie on his back. Then, athletes will be asked to do 90 degrees of knee and hip flexion at the same time. Finally, the athletes is expected to perform slow repetitive knee extension to the point of maximal possible extension. According to Askling et al. and Aspetar protocol, it will be applied 12 repetitions and 3 sets.
  Interventions: Other: Extender Exercise
- Kinesiotaping (Active Comparator): Kinesio taping will be applied to the hamstring muscle in the direction of inhibition with a Y-shaped and 25% tension force.
  Interventions: Other: Kinesiotaping

INTERVENTIONS:
Other: Ballistic Stretching Exercise — It will be applied 4 times per week for 12 weeks.
  Arms: Ballistic Stretching Exercise
Other: Extender Exercise — It will be applied 4 times per week for 12 weeks.
  Arms: Extender Exercise
Other: Kinesiotaping — It will be applied 4 times per week for 12 weeks.
  Arms: Kinesiotaping

SUMMARY:
Low back pain (LBP) is a prevalent issue among adolescent rowers, particularly males aged 14 to 16 years, with a high lifetime prevalence (94%) and point prevalence (65%). One of the mechanisms of lower back pain in rowing athletes is about the elasticity, stiffness and tone of the hamstring muscle.

Current literature shows that stretching exercises, strengthening exercises and kinesiotaping affects hamstring viscoelasticity in various ways. Stretching exercises affect hamstring muscle tone and elasticity, strengthening exercises affect muscle stiffness and kinesiotaping affects muscle tone. While the effects of each of these interventions on viscoelastic properties individually are examined in the literature, studies comparing the effects of changes in viscoelastic properties caused by these interventions on low back pain, athletic disability index and athletic performance in rowers and their superiority among each other are lacking.

The goal of this study is to change the viscoelasticity of the hamstring muscles and examine its effect on low back pain, disability index and athletic performance.

DETAILED DESCRIPTION:
Volunteer male elite rowing athletes between the ages of 14 and 18 who score 3/10 or higher on the Numeric Pain Rating Scale at the time of activity will be included in the study. Signed voluntary consent will be obtained from participants and their legal representatives. Participants will be divided into three groups. Study groups will be as follows: a) ballistic hamstring stretching exercise b) hamstring extender exercise c) kinesiotaping

ELIGIBILITY:
Inclusion Criteria:

* Being between ages 14 and 18 and male gender
* Having been rowing at an elite level for at least one year with a professional team
* Having pain 3/10 or higher on NPRS
* Participating to the study in a voluntary basis.

Exclusion Criteria:

* Having limitation in lower extremity range of motion that limits completion of interventions
* Having a musculoskeletal injury involving the lower extremity in the last 6 months.
* Having undergone a operation in the last 6 months.
* Failing to complete any of interventions.
* Wanting to quit from study.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Frequency of Biceps Femoris Muscle | change from baseline frequency at 12 weeks
  The tones of muscle is described by frequency of muscle or oscillation frequency (Hz). It will be examined by the MyotonPro, Tallinn, Estonia.
Frequency of Semitendinosus Muscle | change from baseline frequency at 12 weeks
  The tones of muscle is described by frequency of muscle or oscillation frequency (Hz). It will be examined by the MyotonPro, Tallinn, Estonia.
Stiffness of Biceps Femoris Muscle | change from baseline frequency at 12 weeks
  Stiffness of muscle is described by reaction to contraction or forces from outside of tissue that may cause the original form to deteriorate. It will be examined by the MyotonPro, Tallinn, Estonia.
Stiffness of Semitendinosus Muscle | change from baseline frequency at 12 weeks
  Stiffness of muscle is described by reaction to contraction or forces from outside of tissue that may cause the original form to deteriorate. It will be examined by the MyotonPro, Tallinn, Estonia.
Numeric Pain Rating Scale (NPRS) | change from baseline pain at the time of activity at 12 weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Standing Long Jump Test (SLJT) | change from baseline performance level at 12 weeks
  It is a horizontal jump test that measures anaerobic performance.
2K-rowing test | change from baseline performance time at 12 weeks
  It is an ergometer test that measures 2,000 meter rowing time and power output as a gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Atakan Sekibağ, MSc, Study Director — Istanbul Nisantasi University
Locations (1):
- İstanbul Nisantasi University, Istanbul, Maslak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noormohammadpour P, Hosseini Khezri A, Farahbakhsh F, Mansournia MA, Smuck M, Kordi R. Reliability and Validity of Athletes Disability Index Questionnaire. Clin J Sport Med. 2018 Mar;28(2):159-167. doi: 10.1097/JSM.0000000000000414. PMID 28107217
- [Background] Ng L, Caneiro JP, Campbell A, Smith A, Burnett A, O'Sullivan P. Cognitive functional approach to manage low back pain in male adolescent rowers: a randomised controlled trial. Br J Sports Med. 2015 Sep;49(17):1125-31. doi: 10.1136/bjsports-2014-093984. Epub 2015 Jan 24. PMID 25618890
- [Background] Yu S, Lin L, Liang H, Lin M, Deng W, Zhan X, Fu X, Liu C. Gender difference in effects of proprioceptive neuromuscular facilitation stretching on flexibility and stiffness of hamstring muscle. Front Physiol. 2022 Jul 22;13:918176. doi: 10.3389/fphys.2022.918176. eCollection 2022. PMID 35941935
- [Background] Almuzaini KS, Fleck SJ. Modification of the standing long jump test enhances ability to predict anaerobic performance. J Strength Cond Res. 2008 Jul;22(4):1265-72. doi: 10.1519/JSC.0b013e3181739838. PMID 18545179
- [Background] Severini G, Holland D, Drumgoole A, Delahunt E, Ditroilo M. Kinematic and electromyographic analysis of the Askling L-Protocol for hamstring training. Scand J Med Sci Sports. 2018 Dec;28(12):2536-2546. doi: 10.1111/sms.13288. Epub 2018 Sep 26. PMID 30171776
- [Background] Askling CM, Tengvar M, Tarassova O, Thorstensson A. Acute hamstring injuries in Swedish elite sprinters and jumpers: a prospective randomised controlled clinical trial comparing two rehabilitation protocols. Br J Sports Med. 2014 Apr;48(7):532-9. doi: 10.1136/bjsports-2013-093214. PMID 24620041
- [Background] van Dyk N, Bahr R, Burnett AF, Whiteley R, Bakken A, Mosler A, Farooq A, Witvrouw E. A comprehensive strength testing protocol offers no clinical value in predicting risk of hamstring injury: a prospective cohort study of 413 professional football players. Br J Sports Med. 2017 Dec;51(23):1695-1702. doi: 10.1136/bjsports-2017-097754. Epub 2017 Jul 29. PMID 28756392
- See also: Hamstring extender exercise — https://www.aspetar.com/journal/viewarticle.aspx?id=440